CLINICAL TRIAL: NCT04758455
Title: P53, Ki67 and Cyclin A Immunohistochemical Staining as Predictors for Wilms' Tumour Aggressiveness and Recurrence
Brief Title: The Use of Immunohistochemical Staining for the Prediction of Wilms Tumour Progression and Recurrence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Ibrahim Atwa, Dr, Mansoura University
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IHS for Wilms tumour relapse
Record Dates: First submitted 2021-02-14; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Wilms Tumor; Relapse; Death
MeSH Terms: conditions — Wilms Tumor; Recurrence; Death | interventions — Genes, p53

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- P53 IHC (Experimental): P53 staining density and intensity will be calculated. To assess P53 density in a semiquantitative way, a score of 0 will be given assigned if less than 5% of tumour cells expressed p53, 1 if 5% to 50% expressed p53 and 2 if more than 50% stained positive for p53. To evaluate P53 intensity, a score of 0 means weak or absent staining, 1 refers to the intermediate intensity and 2 stands for strong intensity.
  Interventions: Diagnostic Test: P53, Ki67 and Cyclin A IHC.
- Ki67 IHC (Experimental): Ki67 proliferation index will be used to detect rapidly proliferating cells which means the percentage of positive Ki67 cells over 5 high power fields. It will be semiquantitatively graded as low, moderate, or high and correlated with histological staging.
  Interventions: Diagnostic Test: P53, Ki67 and Cyclin A IHC.
- Cyclin A IHC (Experimental): Regarding Cyclin A, a standard peroxidase-conjugated streptavidin-biotin labelling was used for visualization, with 3,3 diaminobenzidine as chromogen. Level of cyclin A expression will be classified as absent (-), focal (+), moderate (++) diffuse (+++).
  Interventions: Diagnostic Test: P53, Ki67 and Cyclin A IHC.

INTERVENTIONS:
Diagnostic Test: P53, Ki67 and Cyclin A IHC. — P53, Ki67 and Cyclin A immunohistochemical staining of formalin-fixed paraffin-embedded specimens of Wilms' tumour.

SUMMARY:
Wilms' tumour staging and grading are used to give an idea about the prognosis. Advanced staging, diffuse anaplasia, predominant blastemal elements and lymph node invasion are indicators of poor prognosis. In spite of using the previously mentioned parameters, some tumours which were considered of low risk did not respond to therapy and eventually resulted in mortality. In contrast, other tumours assumed to be of poor prognosis responded dramatically to treatment.

In light of the above, it is crucial to search for predictors of Wilms' tumour prognosis other than tumour staging and grading. Many immunohistochemical (IHC) stains have been studied as prognostic markers for nephroblastoma in literature.

DETAILED DESCRIPTION:
P53 is a tumour suppressor gene, and its mutation is identified in various types of human cancer. P53 protein accumulation in certain tumours is associated with tumour aggressiveness. The role of P53 expression in Wilms' tumour is not clear; however, most studies confirmed its correlation with advanced stages and anaplasia.

Ki67 is a nuclear antigen related to cell proliferation, and high Ki67 proliferation index (PI) is accompanied by tumour aggressiveness, distant metastasis and death. Advanced stages and clinical progression of WT were found to be associated with high Ki67 PI. On the other hand, some authors concluded that it may not be a dependable prognostic marker.

The cyclin-dependent kinases (CDKs) have a role in transitions between cell cycle phases with the need of cyclins association for their activity. IHC assessment of cell cycle proteins has a diagnostic use in histopathology. Correlation between poor prognosis and overexpression of cyclin A was confirmed in different entities of human cancer such as medulloblastoma and ovarian carcinoma. A recent study deduced that cyclin A overexpression may be associated with the poor prognosis of WT.

ELIGIBILITY:
Inclusion Criteria:

* All children presented with Wilms' tumour at the Urology and Nephrology Center, Mansoura University, Mansoura, Egypt from 2000 to 2014.

Exclusion Criteria:

* Preoperative chemotherapy (due to areas of necrosis and haemorrhage hindering immunohistochemical staining).
* Patients with incomplete follow-up data.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-02-14 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
To test the ability of P53, Ki67 and cyclin A to predict Wilms' tumour recurrence and progression. | 2 months
  By correlating P53, Ki67 and cyclin A IHC to tumor stage, histopathology and patients' follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abdelhameed, MSc, Study Chair — Mansoura University; Tamer Helmy, MD, Study Chair — Mansoura University; Ashraf Hafez, MD, Study Director — Mansoura University; Adel Nabeeh, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura Urology and Nephrology Center. Faculty of Medicine, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No